CLINICAL TRIAL: NCT04591405
Title: Phase II/III of Live Attenuated Mumps (F-genotype) Vaccine (Human Diploid Cell, KMB-17) in Healthy Children Aged 5-11
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20190710
Record Dates: First submitted 2020-09-27; First posted 2020-10-19 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Epidemic Parotitis, Mumps
Keywords: Mumps; F-genotype; Live Attenuated Vaccine; Human Diploid Cell
MeSH Terms: conditions — Mumps | interventions — Clinical Trials, Phase II as Topic; Clinical Trials, Phase III as Topic

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Attenuated Mumps vaccine (KMB-17) in phase II and III (Experimental): ≥4.3logCCID50/ml Attenuated Mumps vaccine (KMB-17)[≥4.3 logCCID50/ml] in 360 children (5-11 years old) on 0 day
  Interventions: Biological: Attenuated Mumps vaccine (KMB-17) in phase II and III
- Placebo in phase II (Placebo Comparator): Freeze-dried stabilizer and diluent without mumps virus antigen in 360 children (5-11 years old) on 0 day
  Interventions: Biological: Placebo in phase II
- Attenuated Mumps vaccine (KMB-17) in phase III (Experimental): ≥4.3logCCID50/ml Attenuated Mumps vaccine (KMB-17)[≥4.3 logCCID50/ml] in 5640 children (5-11 years old) on 0 day
  Interventions: Biological: Attenuated Mumps vaccine (KMB-17) in phase III
- Placebo in phase III (Placebo Comparator): Freeze-dried stabilizer and diluent without mumps virus antigen in 5640 children (5-11 years old) on 0 day
  Interventions: Biological: Placebo in phase III

INTERVENTIONS:
Biological: Attenuated Mumps vaccine (KMB-17) in phase II and III — ≥4.3logCCID50/ml Attenuated Mumps vaccine (KMB-17)[≥4.3 logCCID50/ml] in 360 children (5-11 years old) on 0 day
  Arms: Attenuated Mumps vaccine (KMB-17) in phase II and III
Biological: Placebo in phase II — Freeze-dried stabilizer and diluent without mumps virus antigen in 360 children (5-11 years old) on 0 day
  Arms: Placebo in phase II
Biological: Attenuated Mumps vaccine (KMB-17) in phase III — ≥4.3logCCID50/ml Attenuated Mumps vaccine (KMB-17)[≥4.3 logCCID50/ml] in 5640 children (5-11 years old) on 0 day
  Arms: Attenuated Mumps vaccine (KMB-17) in phase III
Biological: Placebo in phase III — Freeze-dried stabilizer and diluent without mumps virus antigen in 5640 children (5-11 years old) on 0 day
  Arms: Placebo in phase III

SUMMARY:
Mumps is an acute infectious respiratory disease caused by the mumps virus (MuV), which occurs mainly in children and adolescents. Its main clinical symptoms were parotid gland suppurative swelling and pain with fever. The pathological changes and harm caused by mumps was not only confined to the parotid gland, on the contrary, the social harm caused by serious complications cannot be ignored. As mumps is a vaccine-preventable infectious disease, vaccination is a fundamental strategy for controlling mumps. So far, there are 13 genotypes of MuV. Based on the analysis of molecular epidemiology, the main epidemic strain of MuV in China was the F genotype. The commonly used vaccine strains represented only a small number of known genotypes, e.g. Jeryl-Lynn (JL) and Rubini strains, which belong to type A, Urabe strain belongs to type B, and L-Zagreb strains belongs to type D. Virus seed of Live Attenuated Mumps Vaccine (Human diploid cell) developed by the institute was SP-A strain, which was the first separation and preparation of the attenuated mumps viruses in China. SP-A belongs to F genotype, which was the domestic epidemic genotype. In addition, the cell substrate prepared for vaccine was human diploid cell (KMB-17 strain), which is much safer to use. The results of phase I and II clinical trials showed that the vaccine possessed good immunogenicity and good antigenic cross-reactivity in infants (8-24 months old).

DETAILED DESCRIPTION:
This study will recruit 12,000 subjects and be divided into two stages. The first stage will evaluate the immunogenicity and safety of F-genotype mumps live attenuated vaccine (human diploid cells) after vaccination in 720 healthy children aged 5-11 years, and explore the detoxification in 144 subjects, who randomly selected from these 720 subjects. The second stage will evaluate the clinical protective efficacy, immunogenicity and safety of F-genotype mumps live attenuated vaccine (human diploid cells) after vaccination in 11280 healthy children aged 5-11 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people aged 5-11 years (including boundary values), both men and women.
* Proven legal identity.
* Participants and parent(s)/legal guardian(s) should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form, and be capable of using thermometers, scales, and filling in diary cards and contact cards as required.
* Participants and parent(s)/legal guardian(s) should be able to communicate well with investigators, understand and comply with the requirements of this trial.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* Contraindications for vaccination.
* History of allergy to vaccines or drugs
* Have a history of mumps disease
* Except for one dose of vaccine containing mumps at the age of 18~24 months before enrollment, any vaccine containing mumps has been vaccinated.
* Any prior administration of attenuated live vaccine in last 15 days;Any prior administration of subunit or inactivated vaccines in last 7 days
* Convulsant,encephalopathy,psychosis or family history of epileptics.
* Those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days.
* For any reason, the spleen was removed partially or completely
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder,it will cause the contraindication of subcutaneous injection
* Suffering from congenital deformity or serious chronic disease(congenital heart disease，Down's syndrome,diabetes,sickle cell anemia,nervous illness,angiocardiopathy,hypertension,bronchitis,pneumonia,asthma,infectious skin diseases)
* Any prior administration of blood products(immunoglobulin etc.) in last 1 month;Any prior administration of immunodepressant, cytotoxic drugs or corticosteroids in last 6 months(except the corticosteroids spray can treat irritability rhinitis or corticosteroids to cure noncomplication acute dermatitis ).
* Receipt of immunosuppressive therapy within 6 months before signing the informed consent form, such as long-term systemic glucocorticoid therapy (with systemic glucocorticoid therapy for more than 2 weeks within 6 months, such as prednisone or similar drugs) ), but local administration (such as ointment, eye drops, inhalation, or nasal spray) is allowed. The local administration should not exceed the dosage recommended in the instructions or have any signs of systemic exposure.
* Any prior administration of other research medicines during the same period.
* Any other situations judged by investigators as not suitable for participating in this study

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11999 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase II: Positive conversion rate of MuV hemagglutination inhibition antibody of Muv Vaccine | 28 day after the vaccination
  To compared the positive conversion rate of MuV hemagglutination inhibition antibody at 28 days after vaccination.
Phase II: Positive conversion rate of MuV neutralization antibody of MuV Vaccine | 28 day after the vaccination
  To compared the positive conversion rate of Muv hemagglutination inhibition antibody at 28 days after vaccination.
Phase III: The protective effect of the MuV vaccine group compared with the placebo group in preventing mumps according with the protocol | within 12 months after vaccination
  To compared the the number of cases of mumps in the vaccine group and the placebo group after 29-day-post injection within 12 months after vaccination

SECONDARY OUTCOMES:
Phase II/III: Adverse reactions/events rate | within 14 days after vaccination
  Occurence of adverse reactions/events within 0-14 days after vaccination
Phase II/III: Adverse reactions/events rate | within 28 days after vaccination
  Occurence of adverse reactions/events within 0-28 days after vaccination
Phase II/III: Serious adverse events rate | within 12 months after vaccination
  Occurence of serious adverse events within 12 months after vaccination
Phase II/III: Positive rate of the hemagglutination inhibition antibody and neutralizing antibody | 28 day after the vaccination
  To compared positive rate of the hemagglutination inhibition antibody and neutralizing antibodies against MuV at 28 days after the vaccination
Phase II/III: The GMT of the hemagglutination inhibition antibody and neutralizing antibody | 28 day after the vaccination
  To compared the GMT of the hemagglutination inhibition antibody and neutralizing antibodies against MuV at 28 days after the vaccination
Phase III: The protective effect of the MuV vaccine group compared with the placebo group in preventing mumps | within 12 months after vaccination
  To compared the the number of cases of mumps in the vaccine group and the placebo group after injection within 12 months after vaccination
Phase III: Positive conversion rate of MuV hemagglutination inhibition antibody of Muv Vaccine | 28 day after the vaccination
  To compared the positive conversion rate of MuV hemagglutination inhibition antibody at 28 days after vaccination.
Phase III: Positive conversion rate of MuV neutralization antibody of MuV Vaccine | 28 day after the vaccination
  To compared the positive conversion rate of Muv hemagglutination inhibition antibody at 28 days after vaccination.
Phase II/III: Positive rate of the hemagglutination inhibition antibody and neutralizing antibody | 12 months after vaccination
  To compared positive rate of the hemagglutination inhibition antibody and neutralizing antibodies against MuV at 12 months after the vaccination
Phase II/III: The GMT of the hemagglutination inhibition antibody and neutralizing antibody | 12 months after vaccination
  To compared the GMT of the hemagglutination inhibition antibody and neutralizing antibodies against MuV at 12 months after the vaccination
Phase II/III: Detoxification | at 3, 7, 14, 28 days after vaccination
  Viral copies in pharyngeal swabs or gargles at 3, 7, 14, 28 days after vaccination were tested by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Qihan Li, Study Chair — Institute of Medical Biology, Chinese Academy of Medical Sciences
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China